CLINICAL TRIAL: NCT02429141
Title: The Ultrasound Guided Periarterial Injection Technique To Axilary Brachial Plexus Block Versus Perineural Multiple InjectionTechnique
Brief Title: Periarterial Injection Versus Multiple Periveural Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North American Institute for Continuing Medical Education (NAICE) (Other)
Responsible Party: Principal Investigator, Catherine Vanderpitt, MD, Catherine Vanderpitte, MD, North American Institute for Continuing Medical Education (NAICE)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAICE-001
Record Dates: First submitted 2015-04-19; First posted 2015-04-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Contusion Wrist or Hand; Crush Injury Wrist or Hand

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- US-guided periarterial techique (Experimental): Axillary brachial plexus block by an ultrasound-guided periarterial technique
  Interventions: Procedure: US-guided periarterial techique
- US-guided multi-injection technique (Experimental): Ultrasound-guided multi-injection perineural technique for axillary brachial plexus
  Interventions: Procedure: US-guided multi-injection technique

INTERVENTIONS:
Procedure: US-guided periarterial techique — The needle will be inserted in the axillary fossa in-plane (cranial to caudal) close to the intersection of the pectoralis and biceps muscles. Two separate injections of local anesthetic will be made deep and superficial to the axillary artery
  Arms: US-guided periarterial techique
Procedure: US-guided multi-injection technique — The median, ulnar and radial nerves will be identified by ultrasound. Local anesthetic will be injected adjacent to each nerve
  Arms: US-guided multi-injection technique

SUMMARY:
In the transarterial technique for axillary brachial plexus block, the axillary artery is intentionally punctured to indicate placement of the needle within the neurovascular sheath; local anesthetic is then injected deep and superficial to the axillary artery.

DETAILED DESCRIPTION:
To lessen the risk for hematoma and intravascular injection, several modifications, such as the multi-injection perineural technique, have become popular. These techniques require a high degree of technical skill and multiple needle passes, and also carry potential for injury. In this study, the investigators will compare an ultrasound-guided equivalent of the transarterial technique (periarterial injections) to a commonly used multi-injection perineural technique.

ELIGIBILITY:
1. Inclusion criteria:

   - Patients (ASA physical status I-III) scheduled to undergo hand or wrist surgery under axillary brachial plexus block
2. Exclusion criteria:

   * Patients with pre-existing neuropathy
   * Patients with allergy to local anesthetics
   * Patients with prior surgery in the ipsilateral axilla
   * Pregnant patients
   * Patients with difficulties in communication

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Block procedure time for the axillary brachial plexus block | time of the block achievement will be recorded up to 15 minutes

SECONDARY OUTCOMES:
Onset of the block | outcome measure will be measured up to 30 minutes a
Time to request pain medication | participants will be followed for 3 days
Block success rate | participants success or block failure within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Admir Hadzic, MD, Study Director — Director
Locations (1):
- Department of Anesthesiology Ziekenhuis Oost-Limburg, Genk, Belgium